CLINICAL TRIAL: NCT00163527
Title: A 24-Week, Double-Blind, Parallel Group, Placebo and Active Controlled Study to Investigate the Efficacy and Safety of Daily Oral Roflumilast Taken With Low Dose Inhaled Corticosteroids in Patients With Chronic Asthma
Brief Title: Efficacy and Safety of Oral Roflumilast Taken With Low Dose Inhaled Corticosteroids in Patients With Asthma (12 to 70 y) (BY217/M2-013)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY217/M2-013
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: Asthma; Roflumilast; Corticosteroids
MeSH Terms: conditions — Asthma | interventions — Roflumilast

INTERVENTIONS:
Drug: Roflumilast

SUMMARY:
Bronchial asthma is among the world's most prevalent diseases. Roflumilast is a novel, orally active, selective enzyme inhibitor (phosphodiesterase 4 inhibitor), which has shown effectiveness in the treatment of asthma.

The aim of the study is to investigate the effect of roflumilast taken orally together with low dose inhaled corticosteroids on lung function. Roflumilast will be administered at one dose level once daily together with inhaled corticosteroids at one dose level twice daily. The study duration consists of a baseline period (2 to 6 weeks) and a treatment period (24 weeks). The study will provide further data on safety, tolerability, and effectiveness of roflumilast.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent
* Diagnosis of persistent chronic bronchial asthma, according to Global Initiative for Asthma (GINA) guidelines
* The patient has been receiving BDP - CFC ≤1000 mcg per day or equivalent for the previous four weeks
* FEV1 between 60 and 90% predicted at visit 1
* No change in asthma treatment within 4 weeks prior to visit 1

Main Exclusion Criteria:

* Patients with poorly controlled asthma defined as requiring a course of oral or parenteral corticosteroids, admission to hospital for asthma (including treatment in an emergency room), or exacerbation of asthma in the four weeks prior to visit 1
* Patients who suffer from seasonal asthma alone or patients who are likely to have a major exacerbation of their asthma due to seasonal effects during the study run-in or treatment period
* A history of lower airway infection in the four weeks prior to visit 1
* A diagnosis of chronic obstructive pulmonary disease (COPD) and/or other relevant lung disease (e.g. cystic fibrosis, bronchiectasis)
* Heavy smoker currently smoking >20 cigarettes per day and/or >10 pack years or the patient is an ex-smoker who has smoked >10 pack years
* Patients using >8 puffs/day relief medication regularly prior to visit 1
* Clinically relevant abnormal laboratory values suggesting an unknown disease and requiring further clinical evaluation
* A diagnosis, treatment or remission of any cancer (other than basal cell carcinoma) within two years prior to visit 1
* Patients with chronic heart failure class III or IV (New York Heart Association)
* Suspected hypersensitivity and/or contraindication to any ingredients of the study medication (roflumilast, BDP, or salbutamol)
* A history of alcoholism or substance abuse within the 12 months prior to visit 1
* Pregnancy or women of childbearing potential who are not using a reliable method of contraception

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2054
Dates: Start 2003-04; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
change in forced expiratory volume in 1 second from baseline to final visit.

SECONDARY OUTCOMES:
change from baseline to each visit for spirometry variables, forced vital capacity, mean expiratory flow, peak expiratory flow
change from baseline to each visit based on diary data variables (asthma symptom scores: daytime, nighttime, and summary, use of rescue medication, diurnal variability)
number of rescue free/symptom free days based on the diary card
area under the curves over the full 24-week trial period for the diary variables
number of exacerbations
time to first exacerbation
change from baseline according to the Asthma Quality of Life Questionnaire (AQLQ).

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (24):
- ALTANA Pharma, Cities in Georgia, Georgia, United States
- ALTANA Pharma, Cities in Austria, Austria
- ALTANA Pharma, Cities in Croatia, Croatia
- ALTANA Pharma, Cities in the Czech Repulik, Czechia
- ALTANA Pharma, Cities in Finland, Finland
- ALTANA Pharma, Cities in France, France
- ALTANA Pharma, Cities in Greece, Greece
- ALTANA Pharma, Cities in Hungary, Hungary
- ALTANA Pharma, Cities in India, India
- ALTANA Pharma, Cities in Ireland, Ireland
- ALTANA Pharma, Cities in Italy, Italy
- ALTANA Pharma, Cities in New Zealand, New Zealand
- ALTANA Pharma, Cities in Norway, Norway
- ALTANA Pharma, Cities in Pakistan, Pakistan
- ALTANA Pharma, Cities in the Philippines, Philippines
- ALTANA Pharma, Cities in Poland, Poland
- ALTANA Pharma, Cities in Portugal, Portugal
- ALTANA Pharma, Cities in the Russian Federation, Russia
- ALTANA Pharma, Sites in Singapore, Singapore
- ALTANA Pharma, Cities in South Africa, South Africa
- ALTANA Pharma, Cities in Spain, Spain
- ALTANA Pharma, Cities in Taiwan, Taiwan
- ALTANA Pharma, Cities in Thailand, Thailand
- ALTANA Pharma, Cities in the United Kindom, United Kingdom

REFERENCES:
- [Derived] Chervinsky P, Meltzer EO, Busse W, Ohta K, Bardin P, Bredenbroker D, Bateman ED. Roflumilast for asthma: Safety findings from a pooled analysis of ten clinical studies. Pulm Pharmacol Ther. 2015 Dec;35 Suppl:S28-34. doi: 10.1016/j.pupt.2015.11.003. Epub 2015 Nov 22. PMID 26612545
- [Derived] Meltzer EO, Chervinsky P, Busse W, Ohta K, Bardin P, Bredenbroker D, Bateman ED. Roflumilast for asthma: Efficacy findings in placebo-controlled studies. Pulm Pharmacol Ther. 2015 Dec;35 Suppl:S20-7. doi: 10.1016/j.pupt.2015.10.006. Epub 2015 Oct 21. PMID 26498386
- See also: BY217-M2-013-RDS-2008-01-21.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4472&filename=BY217-M2-013-RDS-2008-01-21.pdf